CLINICAL TRIAL: NCT02379169
Title: Effects of Sea Buckthorn Oil and Lutein on Eye Health
Acronym: SBEYE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Turku University Hospital (Other Government)
Collaborators: Aromtech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SBEYE
Record Dates: First submitted 2014-11-07; First posted 2015-03-04 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2014-11

CONDITIONS: Risk Factors for Age Related Macular Degeneration
Keywords: macular pigment optical density, age related macular degeneration, dry eye, vision
MeSH Terms: conditions — Macular Degeneration; Dry Eye Syndromes | interventions — Lutein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sea buckthorn & lutein (Experimental): Sea buckthorn oil complemented with lutein. Dose: 2 g/day as capsules taken twice/day for 6 months
  Interventions: Dietary Supplement: Sea buckthorn oil & lutein
- Placebo (Placebo Comparator): Triglycerides of medium-chain fatty acids. Dose: 2 g/day as capsules taken twice/day for 6 months
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Sea buckthorn oil & lutein — Standardised sea buckthorn seed and pulp oil complemented with lutein
  Arms: Sea buckthorn & lutein
Dietary Supplement: Placebo — Triglycerides of medium chain fatty acids
  Arms: Placebo

SUMMARY:
Low macular pigment optical density has been associated with increased risk of age-related macular degeneration, an important cause of vision problems in the elderly population. Dry eye is multifactorial disease of tears and the ocular surface associated with symptoms of dryness, grittiness, burning and redness of eyes. The risk of dry eye increases with age. The aim is to investigate the effects of sea buckthorn oil complemented with lutein on eye health, specifically on the macula.

ELIGIBILITY:
Inclusion Criteria:

- macular pigment optical density equal to or less than 0,40 OD

Exclusion Criteria:

* diabetic retinopathy
* macular changes associated with high blood pressure
* signs of macular degeneration: classes 2, 3 and 4 according to the Rotterdam study (Mol Vis 2012: 657-74)
* severe eye diseases, exluding cataract. The intervention will begina after surgery and recovery from cataract

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-02 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Change in macular pigment optical density from baseline to 6 mo | 0 mo, 3 mo, 6 mo
  measurement of macular pigment optical density

SECONDARY OUTCOMES:
Change in symptoms of dry eye from baseline to 6 mo | 0 months, 3 months, 6 months
  questionnaires, symptom logbook
Change in serum lipids (Triglycerides, HDL-cholesterol, LDL-cholesterol, total cholesterol) from baseline to 6 mo | 0 months, 6 months
  analysis from serum samples
Change in serum markers of inflammation (hs-CRP) from baseline to 6 mo | 0 months, 6 months
  analysis from serum samples
Change in circulating aminotransferases (ALAT, ASAT) from baseline to 6 mo | 0 months, 6 months
  analysis from plasma samples
Change in contrast sensitivity from baseline to 6 mo | 0 mo, 3 mo, 6 mo
  analysis of contrast sensitivity
Change in vision aquity from baseline to 6 mo | 0 mo, 3 mo, 6 mo
  ETDRS chart
Change in vision functioning from baseline to 6 mo | 0 mo, 3 mo, 6 mo
  questionnaire
Change in tear film osmolarity from baseline to 6 mo | 0 mo, 3 mo, 6 mo
  measurement of tear film osmolarity

OTHER OUTCOMES:
Change in serum markers of sea buckthorn oil and lutein intake | 0 months, 6 months
  analysis from serum samples